CLINICAL TRIAL: NCT05132530
Title: The Effect of Yoga Training on Adolescents on Psychological Resilience and Stress Management
Acronym: Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sinem Dağ, SENİOR INSTRUCTOR, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ETK00-2021-0187; Emine Öksüz (Other: sağlık bilimleri üniversitesi)
Record Dates: First submitted 2021-10-15; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Adolescent
Keywords: Yoga; Adolescent; Stress
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Gruop (Experimental): Experimental: İntervention Group
  Yoga practice will be practiced 2 days a week for 10 weeks.
  Interventions: Behavioral: yoga
- Control Group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: yoga — yoga practice will be done two days a week for 10 weeks.
  Arms: Intervention Gruop

SUMMARY:
Adolescents may experience daily difficulties in family and peer relationships, due to school and exams. These troubles are disturbing and obstructive events that can cause the stress that people usually encounter in their environmental interactions. It can negatively affect people's mental and physical health. It is stated that yoga regulates the nervous system and physiological functioning of the body, provides physical fitness and improves psychological well-being. However, it calms the soul and supports mental health. In this study, it was aimed to determine the effect of yoga training applied to 13-16 years old adolescents for 10 weeks on their psychological resilience and coping with stress.

DETAILED DESCRIPTION:
Adolescence is the period of transition from childhood to adulthood in which rapid growth, development and maturation occur in terms of biochemical, physical, social and spiritual aspects. It is thought that yoga practice will be beneficial for adolescents to spend this risky period in a healthy way, to cope with psychological resilience and stress, and to practice yoga as a lifestyle in other periods is thought to be effective. Adolescents living in the Famagusta region, aged 13-16, willing to participate in the research and applying for yoga groups, who meet the research criteria. After the applications, the adolescents who meet the research criteria and volunteer to participate in the research will be listed and the adolescents in the list will be randomly selected into the study and control groups using the random numbers table. In the study, data will be collected with a data collection form consisting of two parts: "Descriptive Characteristics Form", "Child and Youth Psychological Resilience Scale, and Adolescent Coping Scale". In the study, there will be two groups, the study and the control, selected by randomization. Adolescents who meet the research criteria will be informed about the research in the conference hall of Famagusta Development Academy. Informed (voluntary) consent forms will be signed by the adolescents and parents who agree to participate in the study. A data collection form will be applied to all adolescents participating in the study. In the research, yoga groups will be formed by determining the appropriate day and time for the adolescents in the study group. Adolescents in the study group will have 60 minutes of yoga practice twice a week for 10 weeks. Yoga practice will be performed by the researcher in the dance hall of Famagusta Development Academy. After the 10-week yoga training period is over, it will be filled by the adolescents in the last yoga class. No intervention will be made in the control group. At the end of 10 weeks, questionnaires will be applied to the control group again.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the research,
* Open to communication,
* between the ages of 13-16
* Diagnosed musculoskeletal disease, without advanced heart disease,
* Not doing regular exercise and yoga,

Exclusion Criteria:

* Those who do not agree to participate in the research,
* Unable to communicate
* under the age of 13, over the age of 16,
* Those with diagnosed musculoskeletal disease, advanced heart disease,
* Regular exercise and yoga,

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Among adolescent girls 13-16 years old
Enrollment: 60 (Estimated)
Dates: Start 2021-12-08 (Estimated); Primary Completion 2021-12-08 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Child and Youth Psychological Resilience Scale | 10 weeks
  The short formula of the scale consisting of 12 items was made by Ungar, Liebenberg, and LeBlanc (2013) (Liebenberg et al., 2013). The popular heights of children and young youth are seen as .39 and .84 from the inside. According to the five-point Likert scale in the scale, it is answered as "Describes me (5)" and "Does not describe me at all (1)". A high score indicates high robustness. The Turkish adaptation of the scale and its reliability-validity study were performed by Arslan (2015). A minimum of 12 points and a maximum of 60 points can be obtained from the scale. High score values indicate a high level of resilience.The factor loads of twelve items of the Child and Adolescent Resilience Scale ranged from .54 to .81. This situation is important in terms of showing the high level of representativeness power of the items in the scale.
Coping Scale for Adolescents | 10 weeks
  The validity and reliability of the Turkish version of the Coping Scale for Adolescents developed by Spirito, Stark and Williams (1988) was determined by Bedel et al. He did it in 2014.The adolescent form used ten coping strategies (social distancing, distraction, wishful thinking, cognitive restructuring, It consists of 11 items measuring social support, problem solving, self-criticism, emotion regulation, withdrawal, and blaming others. Ratings are made on a four-point scale: Never (0), Sometimes (1), Often (2), and Always (3). Scale scoring, Active Coping: 3, 6, 8, 10 Avoidant Coping: 1, 2, 9, 11 Negative Coping: 4, 5, 7. For Scale Evaluation, Each subscale score is obtained by summing the related items in order. The possible scores range from 0-12 for Active coping and Avoidant coping, and 0-9 for Negative coping.
  Higher scores indicate that the relevant coping approach is used more frequently.

CONTACTS AND LOCATIONS:
Overall Officials: sinem dağ, phd, Principal Investigator — recruiting
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Yoga in school settings: a research review — https://pubmed.ncbi.nlm.nih.gov/26919395/
- See also: A yoga program for cognitive enhancement — https://pubmed.ncbi.nlm.nih.gov/28783749/
- See also: INDIVIDUALIZED YOGA FOR REDUCING DEPRESSION AND ANXIETY, AND IMPROVING WELL-BEING: A RANDOMIZED CONTROLLED TRIAL — https://pubmed.ncbi.nlm.nih.gov/27030303/
- See also: Systematic Review of Yoga Interventions for Anxiety Reduction Among Children and Adolescents — https://pubmed.ncbi.nlm.nih.gov/26565100/